CLINICAL TRIAL: NCT02789514
Title: A Survey of the Indications for Esophagogastroduodenoscopy (EGD) in Children's Hospital of Fudan University
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ying HUANG, The director of gastroenterology of Children's Hospital of Fudan University, Children's Hospital of Fudan University
Other Study IDs: fudanU-E1
Record Dates: First submitted 2016-05-19; First posted 2016-06-03 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Digestive System Abnormalities
Keywords: esophagogastroduodenoscopy; paediatric
MeSH Terms: conditions — Digestive System Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- children: Investigators give observation to the patients who need esophagogastroduodenoscopic procedures.

SUMMARY:
Esophagogastroduodenoscopy (EGD) become more and more common in diagnosing gastroenterology diseases. The investigators want to find which symptoms can support for positive endoscopic findings.

DETAILED DESCRIPTION:
Esophagogastroduodenoscopy (EGD) become more and more common in diagnosing gastroenterology diseases. And there are indications for EGD. Here, investigators want to find which symptoms can strongly support for positive endoscopy findings. So, investigators design the study to record the symptoms in detail and diagnosis, and then analysis symptoms and the rate of endoscopic findings.

ELIGIBILITY:
Inclusion Criteria:

* All of the patients need esophagogastroduodenoscopic procedures

Exclusion Criteria:

* None

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All of the patients need esophagogastroduodenoscopic procedures
Sampling Method: Non-Probability Sample
Enrollment: 1303 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Questionnaires about the indications for esophagogastroduodenoscopic procedures were collected | May, 2016-August, 2016
  The content of questionnaire include the symptoms which prompt for the esophagogastroduodenoscopic procedure, and the diagnosis. Then investigators will analysis the relationship between symptom and diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Huang, doctor, Study Director — Children's Hospital of Fudan University

IPD SHARING:
Plan to Share IPD: Undecided